CLINICAL TRIAL: NCT05161403
Title: The Efficacy of Hyaluronic Acid and Honey in Healing of Multiple Extraction Sockets of Primary Teeth Compared to Saline in a Group of Egyptian Children
Brief Title: The Efficacy of Hyaluronic Acid and Honey in Healing of Multiple Extraction Sockets of Primary Teeth Compared to Saline
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Anas Rahima, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: wound healing on pediatric
Record Dates: First submitted 2021-10-26; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-11

CONDITIONS: Wound Heal
MeSH Terms: interventions — Hyaluronic Acid; Honey

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Masking Description: Neither the operator nor the patients could be blinded due to the nature of the study, but the statistician will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hyaluronic acid. (Active Comparator): 1mm layer of hyaluronic acid on a piece of gauze will be applied directly to the sockets wound for 45 minutes at baseline and on the third & seventh day after extraction of teeth.
  Interventions: Drug: Hyaluronic acid; Dietary Supplement: honey
- Honey (Active Comparator): 1mm layer of Honey on a piece of gauze will be applied directly to the sockets wound for 45 minutes at baseline and on the third & seventh day after extraction of teeth.
  Interventions: Drug: Hyaluronic acid; Dietary Supplement: honey
- Saline (Placebo Comparator): a piece of gauze moistened with normal saline will be applied directly to the sockets wound for 45 minutes at baseline and on the third & seventh day after extraction of teeth.
  Interventions: Drug: Hyaluronic acid; Dietary Supplement: honey

INTERVENTIONS:
Drug: Hyaluronic acid — Wound healing is still a clinical challenge especially in patients who undergo several tooth extractions under general anesthesia or those undergoing major surgeries or those with systemic conditions that disrupt the wound healing process.
  use of this natural substance is a simple and cost-effective technique and is easily tolerated by children.
Dietary Supplement: honey — Wound healing is still a clinical challenge especially in patients who undergo several tooth extractions under general anesthesia or those undergoing major surgeries or those with systemic conditions that disrupt the wound healing process.
  Use of this natural substance is a simple and cost-effective technique and is easily tolerated by children.

SUMMARY:
This study aims to evaluate the effect of hyaluronic acid and honey compared to saline in healing of multiple extraction sockets of primary teeth in a group of children aging from Two to Seven years old.

DETAILED DESCRIPTION:
A dental extraction is one of the most unpleasant experiences in children, especially for those who have undergone traumatic experiences, and this is likely to reduce future visits to the dental clinic if the treatment is not managed properly.

Alveolar osteitis is one of the most common complications following dental extraction. It is considered one of the most studied complications in dentistry, and many risk factors contribute to its occurrence including being a female, young age, tobacco use, difficult or traumatic extractions, pre-existing infection, and use of vasoconstrictor in local anesthesia. Alveolar osteitis occurs during the first three days following the day of extraction, so that the socket is devoid of the blood clot, resulting in the exposure of the bare alveolar bone.

Many medicines were and are still used in treating wounds, but they are somewhat expensive.

ELIGIBILITY:
Inclusion Criteria:

* • Age: from Two to Seven years old age.

  * Both genders.
  * Children with badly decayed multiple primary teeth beyond repair.
  * Treated under general anesthesia.

Exclusion Criteria:

* • History of systemic disease.

  * Allergy to honey.
  * Repeatedly used honey during the previous 6 month period.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Estimated)
Dates: Start 2022-02-22 (Estimated); Primary Completion 2023-09-04 (Estimated); Study Completion 2023-09-04 (Estimated)

PRIMARY OUTCOMES:
Wound healing size in length and width | After one week will be calculated the size (lentgh and width) of socket
  There is only one outcome (wound healing)
  • Multiple measurements (Digital caliper, color, palpation, presence of pus, gingival margin status).
  1. Digital caliper: a device used to calculate the size of the socket (width and length) buccolingual in mesiodistal with measurement of mm.
  2. Color: normal (pinkish gingiva) Up normal (reddish gingiva)
  3. Palpation: if there is bleeding or not.
  4. Presence of pus: yes or no
  5. Gingival margin: epithelization (yes or no)

REFERENCES:
- [Result] Naaman R, El-Housseiny AA, Alamoudi N, Helal N, Sahhaf R. Reliability and Validity of the Arabic Version of a Questionnaire Assessing Pain, Discomfort and Related Jaw Function Impairment after Extraction of Primary Teeth in Children. Dent J (Basel). 2020 Oct 19;8(4):120. doi: 10.3390/dj8040120. PMID 33086538
- [Result] Iacopetti I, Perazzi A, Martinello T, Gemignani F, Patruno M. Hyaluronic acid, Manuka honey and Acemannan gel: Wound-specific applications for skin lesions. Res Vet Sci. 2020 Apr;129:82-89. doi: 10.1016/j.rvsc.2020.01.009. Epub 2020 Jan 11. PMID 31954318
- [Result] Maria de Souza G, Elias GM, Pereira de Andrade PF, Andrade Sales KN, Galvao EL, Moreira Falci SG. The Effectiveness of Hyaluronic Acid in Controlling Pain, Edema, and Trismus After Extraction of Third Molars: Systematic Review and Meta-Analysis. J Oral Maxillofac Surg. 2020 Dec;78(12):2154.e1-2154.e12. doi: 10.1016/j.joms.2020.07.005. Epub 2020 Jul 14. PMID 32771444
- [Result] Mokhtari S, Sanati I, Abdolahy S, Hosseini Z. Evaluation of the effect of honey on the healing of tooth extraction wounds in 4- to 9-year-old children. Niger J Clin Pract. 2019 Oct;22(10):1328-1334. doi: 10.4103/njcp.njcp_102_19. PMID 31607720
- [Result] Jaffe HW, Sweeney HM, Weinstein RA, Kabins SA, Nathan C, Cohen S. Structural and phenotypic varieties of gentamicin resistance plasmids in hospital strains of Staphylococcus aureus and coagulase-negative staphylococci. Antimicrob Agents Chemother. 1982 May;21(5):773-9. doi: 10.1128/AAC.21.5.773. PMID 7103456